CLINICAL TRIAL: NCT04857060
Title: Meeting the Challenges of COVID-19 by Expanding the Reach of Palliative Care: Proactive Advance Care Planning With Videos for the Elderly and All Patients With Dementia
Brief Title: Palliative Care Educator
Acronym: VIDEO-PCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-41482; 1R01AG072911-01 (NIH)
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Advance Care Planning; Palliative Care; Alzheimer's Disease and Related Dementias; Doctor-patient Communication; Video Decision Aids
Keywords: video decision aid; palliative care educator
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Subjects in this arm do not meet with ACP Educator during their index hospitalization.
- ACP Educator led, video assisted discussion (Experimental): For hospitalized patients identified by a defined EHR algorithm, an ACP Educator will meet with the patient in the hospital to provide primary palliative care services such as goals-of-care conversations and clinician communication by leveraging certified video decision aids.
  Interventions: Behavioral: ACP Educator led, video assisted discussion

INTERVENTIONS:
Behavioral: ACP Educator led, video assisted discussion — For hospitalized patients identified by a defined EHR algorithm, an ACP Educator will meet with the patient in the hospital to provide primary palliative care services such as goals-of-care conversations and clinician communication by leveraging certified video decision aids.
  Arms: ACP Educator led, video assisted discussion

SUMMARY:
The investigators propose to conduct a stepped wedge cluster randomized trial of an advance care planning (ACP) educator-led intervention among hospitalized patients aged 65 and over, or any patient with Alzheimer's Disease and Related Dementias (ADRD) and their proxy decision-makers in the ward and ICU settings of two major hospitals: Boston Medical Center and North Shore University Hospital in New York. Patient outcomes will be abstracted from electronic health records with Natural Language Processing. The effectiveness of the intervention will be evaluated by comparing the following outcomes among 9,000 hospitalized patients (Aim 1): ACP documentation; preferences for resuscitation; palliative care consults; and, hospice use. The investigators will characterize caregiver-centered outcomes of patients with ADRD, including (Aim 2): (1) knowledge, (2) confidence in future care, (3) communication satisfaction, and (4) decisional certainty in 600 caregivers of patients with ADRD admitted to the hospital. COVID-19 poses a unique dilemma for older Americans and patients with ADRD and their caregivers, who must balance their desire to live against the risk of a lonely and potentially traumatic hospital death. Video decision support is a practical, evidence-based, and innovative approach to assist patients facing such choices. If proven effective, this innovative care model can be immediately deployed across the country to improve the quality of care for millions of Americans.

DETAILED DESCRIPTION:
The majority of patients aged 65 or over, and patients with Alzheimer's Disease and Related Dementias (ADRD), have never communicated their preferences to clinicians or completed advance care planning (ACP) documents. Palliative care has the potential to improve ADRD care, improve patient-clinician communication and patient-centered outcomes, while decreasing unwanted burdensome treatments and improving care at the end of life. The novel Coronavirus Disease 2019 (COVID-19) has acutely escalated the importance of integrating ACP and palliative care services into medical care. The default response to critical illness for patients with ADRD (and all others) is intubation, mechanical ventilation, and aggressive care despite having no change in mortality outcome. ADRD patients and their caregivers may prefer to avoid these interventions.

To address these gaps, the investigators have developed a COVID-19 ACP Educator-led, video-assisted palliative care intervention to improve patient-clinician communication, increase ACP documentation, and lead to more patient-centered care at the end of life. The investigators will identify all hospitalized patients aged 65 and older, and any patient with ADRD, and then an ACP Educator will proactively proceed with primary palliative care services of ACP, leveraging certified video decision aids developed by the research team. This will be considered the standard of care for all patients meeting eligibility criteria. The ACP Educator to be tested in this proposal represents a new role and proactive function for the palliative care team. The ACP Educator will work with older patients or patients with ADRD and proxy decision-makers to learn about and document patients' wishes.

ELIGIBILITY:
Inclusion Criteria: Aim 1

* Inpatient at study sites
* Age 65 and older

Inclusion Criteria: Aim 2 (Caregiver Survey)

* Age 18 and older
* Designated caregiver of inpatient identified in Aim 1 who are diagnosed with Alzheimer's Disease and Related Dementias or other cognitive impairments
* English or Spanish speaking

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11174 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Paasche-Orlow, MD, MPH, Principal Investigator — Tufts Medical Center
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Northshore University Hospital, Manhasset, New York

IPD SHARING:
Plan to Share IPD: Yes
The phenotypic data associated with enrolled participants will be shared by depositing these data in the Open Science Framework data repository. Additional data documentation and de-identified IPD including demographics, diagnoses, and outcomes will be deposited. Resources such as study protocols and statistical analysis codes will also be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Outcome data will be deposited into Open Science Framework repository as soon as possible but no later than within one year of the completion of the funded project period for the parent award or upon acceptance of the data for publication, or public disclosure of a submitted patent application, whichever is earlier. Data will remain available for a period of 5 years.
Access Criteria: Data and supporting information will be shared with investigators working in accordance to guidelines set by the data repository. Meta-analysis data and associated phenotypic data, along with data content, format, and organization, will be made available to investigators through the Open Science Framework data repository.

REFERENCES:
- [Derived] Zupanc SN, Quintiliani LM, LeClair AM, Paasche-Orlow MK, Volandes A, Penumarthy A, Henault L, Itty JE, Davis AD, Lakin JR. The Sowers of Seeds: A Qualitative Analysis of the Role of Palliative Care Educators in Facilitating Goals-of-Care Conversations and Palliative Care Referrals. Am J Hosp Palliat Care. 2025 Aug;42(8):761-768. doi: 10.1177/10499091241267917. Epub 2024 Aug 28. PMID 39196855
- [Derived] Volandes AE, Zupanc SN, Lakin JR, Cabral HJ, Burns EA, Carney MT, Lopez S, Itty J, Emmert K, Martin NJ, Cole T, Dobie A, Cucinotta T, Joel M, Caruso LB, Henault L, Dugas JN, Astone K, Winter M, Wang N, Davis AD, Garde C, Rodriguez PM, El-Jawahri A, Moseley ET, Das S, Sciacca K, Ramirez AM, Gromova V, Lambert S, Sanghani S, Lindvall C, Paasche-Orlow MK. Video Intervention and Goals-of-Care Documentation in Hospitalized Older Adults: The VIDEO-PCE Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2332556. doi: 10.1001/jamanetworkopen.2023.32556. PMID 37695586
- [Derived] Lakin JR, Zupanc SN, Lindvall C, Moseley ET, Das S, Sciacca K, Cabral HJ, Burns EA, Carney MT, Itty J, Lopez S, Emmert K, Martin NJ, Lambert S, Polo J, Sanghani S, Dugas JN, Gomez M, Winter MR, Wang N, Gabry-Kalikow S, Dobie A, Amshoff M, Cucinotta T, Joel M, Caruso LB, Ramirez AM, Salerno K, Ogunneye Q, Henault L, Davis AD, Volandes A, Paasche-Orlow MK. Study protocol for Video Images about Decisions to Improve Ethical Outcomes with Palliative Care Educators (VIDEO-PCE): a pragmatic stepped wedge cluster randomised trial of older patients admitted to the hospital. BMJ Open. 2022 Jul 25;12(7):e065236. doi: 10.1136/bmjopen-2022-065236. PMID 35879001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included patients aged 65 years or older and their caregivers admitted to 1 of 14 units at two urban hospitals in New York and Boston from July 1, 2021, to October 31, 2022.
Pre-assignment Details: Of the 11,174 participants, 6,201 participants were randomized into the intervention.
Units Other Than Participants: Inpatient unit
Groups:
- Step 0: 2 Months Usual Care Then 14 Months ACP Educator Led, Video Assisted Discussion; Step 1: 4 Months Usual Care, Then 10 Months ACP Educator Led, Video Assisted Discussion; Step 2: 6 Months Usual Care, Then 8 Months ACP Educator Led, Video Assisted Discussion; Step 3: 8 Months Usual Care, Then 6 Months ACP Educator Led, Video Assisted Discussion; Step 4: 10 Months Usual Care, Then 4 Months ACP Educator Led, Video Assisted Discussion; Step 5: 12 Months Usual Care, Then 2 Months ACP Educator Led, Video Assisted Discussion; Step 6: 14 Months Usual Care, Then 0 Months ACP Educator Led, Video Assisted Discussion: For hospitalized patients identified by a defined EHR algorithm, an ACP Educator will meet with the patient in the hospital to provide primary palliative care services such as goals-of-care conversations and clinician communication by leveraging certified video decision aids.
  ACP Educator led, video assisted discussion: For hospitalized patients identified by a defined EHR algorithm, an ACP Educator will meet with the patient in the hospital to provide primary palliative care services such as goals-of-care conversations and clinician communication by leveraging certified video decision aids.
Period: Control: Usual Care (Patients)
Arm/Group | Step 0: 2 Months Usual Care Then 14 Months ACP Educator Led, Video Assisted Discussion | Step 1: 4 Months Usual Care, Then 10 Months ACP Educator Led, Video Assisted Discussion | Step 2: 6 Months Usual Care, Then 8 Months ACP Educator Led, Video Assisted Discussion | Step 3: 8 Months Usual Care, Then 6 Months ACP Educator Led, Video Assisted Discussion | Step 4: 10 Months Usual Care, Then 4 Months ACP Educator Led, Video Assisted Discussion | Step 5: 12 Months Usual Care, Then 2 Months ACP Educator Led, Video Assisted Discussion | Step 6: 14 Months Usual Care, Then 0 Months ACP Educator Led, Video Assisted Discussion
Started (Step 0: There are 14 units total. All units start in the control group and then receive the intervention after 2 months of usual care.) | 1698; 2 Inpatient unit | 1190; 2 Inpatient unit | 853; 2 Inpatient unit | 543; 2 Inpatient unit | 357; 2 Inpatient unit | 88; 2 Inpatient unit | 50; 2 Inpatient unit
Completed | 1698; 2 Inpatient unit | 1190; 2 Inpatient unit | 853; 2 Inpatient unit | 543; 2 Inpatient unit | 357; 2 Inpatient unit | 88; 2 Inpatient unit | 50; 2 Inpatient unit
Not Completed | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit
Period: Intervention:Video Discussion (Patients)
Arm/Group | Step 0: 2 Months Usual Care Then 14 Months ACP Educator Led, Video Assisted Discussion | Step 1: 4 Months Usual Care, Then 10 Months ACP Educator Led, Video Assisted Discussion | Step 2: 6 Months Usual Care, Then 8 Months ACP Educator Led, Video Assisted Discussion | Step 3: 8 Months Usual Care, Then 6 Months ACP Educator Led, Video Assisted Discussion | Step 4: 10 Months Usual Care, Then 4 Months ACP Educator Led, Video Assisted Discussion | Step 5: 12 Months Usual Care, Then 2 Months ACP Educator Led, Video Assisted Discussion | Step 6: 14 Months Usual Care, Then 0 Months ACP Educator Led, Video Assisted Discussion
Started | 263; 2 Inpatient unit | 495; 2 Inpatient unit | 650; 2 Inpatient unit | 979; 2 Inpatient unit | 1178; 2 Inpatient unit | 1212; 2 Inpatient unit | 1246; 2 Inpatient unit
Completed | 263; 2 Inpatient unit | 495; 2 Inpatient unit | 650; 2 Inpatient unit | 979; 2 Inpatient unit | 1178; 2 Inpatient unit | 1212; 2 Inpatient unit | 1246; 2 Inpatient unit
Not Completed | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit
Period: Control: Usual Care (Caregiver)
Arm/Group | Step 0: 2 Months Usual Care Then 14 Months ACP Educator Led, Video Assisted Discussion | Step 1: 4 Months Usual Care, Then 10 Months ACP Educator Led, Video Assisted Discussion | Step 2: 6 Months Usual Care, Then 8 Months ACP Educator Led, Video Assisted Discussion | Step 3: 8 Months Usual Care, Then 6 Months ACP Educator Led, Video Assisted Discussion | Step 4: 10 Months Usual Care, Then 4 Months ACP Educator Led, Video Assisted Discussion | Step 5: 12 Months Usual Care, Then 2 Months ACP Educator Led, Video Assisted Discussion | Step 6: 14 Months Usual Care, Then 0 Months ACP Educator Led, Video Assisted Discussion
Started | 4; 2 Inpatient unit | 28; 2 Inpatient unit | 39; 2 Inpatient unit | 33; 2 Inpatient unit | 27; 2 Inpatient unit | 31; 2 Inpatient unit | 32; 2 Inpatient unit
Completed | 4; 2 Inpatient unit | 28; 2 Inpatient unit | 39; 2 Inpatient unit | 33; 2 Inpatient unit | 27; 2 Inpatient unit | 31; 2 Inpatient unit | 32; 2 Inpatient unit
Not Completed | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit
Period: Intervention:Video Discussion(Caregiver)
Arm/Group | Step 0: 2 Months Usual Care Then 14 Months ACP Educator Led, Video Assisted Discussion | Step 1: 4 Months Usual Care, Then 10 Months ACP Educator Led, Video Assisted Discussion | Step 2: 6 Months Usual Care, Then 8 Months ACP Educator Led, Video Assisted Discussion | Step 3: 8 Months Usual Care, Then 6 Months ACP Educator Led, Video Assisted Discussion | Step 4: 10 Months Usual Care, Then 4 Months ACP Educator Led, Video Assisted Discussion | Step 5: 12 Months Usual Care, Then 2 Months ACP Educator Led, Video Assisted Discussion | Step 6: 14 Months Usual Care, Then 0 Months ACP Educator Led, Video Assisted Discussion
Started | 8; 2 Inpatient unit | 18; 2 Inpatient unit | 15; 2 Inpatient unit | 34; 2 Inpatient unit | 30; 2 Inpatient unit | 19; 2 Inpatient unit | 54; 2 Inpatient unit
Completed | 8; 2 Inpatient unit | 18; 2 Inpatient unit | 15; 2 Inpatient unit | 34; 2 Inpatient unit | 30; 2 Inpatient unit | 19; 2 Inpatient unit | 54; 2 Inpatient unit
Not Completed | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit | 0; 0 Inpatient unit

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACP Educator Led, Video Assisted Discussion | Usual Care | Total
Number analyzed (Participants) | 6208 | 4985 | 11193
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The row population differs from the overall to show the difference between patients and caregivers.
  years
    Patient: number analyzed (Participants) | 6023 | 4779 | 10802
    Patient | 78 (8) | 78 (8) | 78 (8)
    Caregivers: number analyzed (Participants) | 178 | 194 | 372
    Caregivers | 57 (13) | 57 (13) | 57 (13)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The rows are different to represent both caregivers and patients included in the analysis
  Participants
    Patients: number analyzed (Participants) | 6023 | 4779 | 10802
    Patients: Female | 2888 | 2335 | 5223
    Patients: Male | 3135 | 2444 | 5579
    Patients: Unknown or not reported | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 178 | 194 | 372
    Caregivers: Female | 119 | 129 | 248
    Caregivers: Male | 52 | 64 | 116
    Caregivers: Unknown or not reported | 7 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The rows differ to represent patient and caregiver data
  Participants
    Patients: number analyzed (Participants) | 6023 | 4779 | 10802
    Patients: Hispanic or Latino | 548 | 451 | 999
    Patients: Not Hispanic or Latino | 5337 | 4200 | 9537
    Patients: Unknown or Not Reported | 138 | 128 | 266
    Caregivers: number analyzed (Participants) | 178 | 194 | 372
    Caregivers: Hispanic or Latino | 23 | 18 | 41
    Caregivers: Not Hispanic or Latino | 149 | 171 | 320
    Caregivers: Unknown or Not Reported | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The row differs to show patient and caregiver data collected
  Participants
    Patients: number analyzed (Participants) | 6023 | 4779 | 10802
    Patients: American Indian or Alaska Native | 16 | 14 | 30
    Patients: Asian | 509 | 386 | 895
    Patients: Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
    Patients: Black or African American | 1376 | 1125 | 2501
    Patients: White | 3113 | 2483 | 5596
    Patients: More than one race | 617 | 454 | 1071
    Patients: Unknown or Not Reported | 390 | 314 | 704
    Caregivers: number analyzed (Participants) | 178 | 194 | 372
    Caregivers: American Indian or Alaska Native | 2 | 1 | 3
    Caregivers: Asian | 9 | 5 | 14
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers: Black or African American | 61 | 63 | 124
    Caregivers: White | 84 | 110 | 194
    Caregivers: More than one race | 3 | 3 | 6
    Caregivers: Unknown or Not Reported | 19 | 12 | 31
Region of Enrollment [Number; unit: participants]
  United States | 6208 | 4985 | 11193
Language [Number; unit: participants] — Population: The rows differ to represent show the difference in caregiver and participant data
  participants
    English (Patient): number analyzed (Participants) | 6023 | 4779 | 10802
    English (Patient) | 4909 | 3864 | 8773
    Spanish (Patient): number analyzed (Participants) | 6023 | 4779 | 10802
    Spanish (Patient) | 352 | 315 | 667
    Other (Patient): number analyzed (Participants) | 6023 | 4779 | 10802
    Other (Patient) | 707 | 548 | 1255
    Unknown or missing (Patient): number analyzed (Participants) | 6023 | 4779 | 10802
    Unknown or missing (Patient) | 55 | 52 | 107
    English (Caregiver): number analyzed (Participants) | 178 | 194 | 372
    English (Caregiver) | 172 | 190 | 362
    Spanish (Caregiver): number analyzed (Participants) | 178 | 194 | 372
    Spanish (Caregiver) | 6 | 4 | 10
    Other (Caregiver): number analyzed (Participants) | 178 | 194 | 372
    Other (Caregiver) | 0 | 0 | 0
    Unknown or missing (Caregiver): number analyzed (Participants) | 178 | 194 | 372
    Unknown or missing (Caregiver) | 0 | 0 | 0
Alzheimer's disease and related dementias diagnosis [Number; unit: participants] — ADRD Diagnosis was only collected for patients Population: The row population differs from the overall since data only from patients was collected about ADRD diagnosis, and not from caregivers.
  participants
    Yes: number analyzed (Participants) | 6023 | 4779 | 10802
    Yes | 681 | 570 | 1251
    No: number analyzed (Participants) | 6023 | 4779 | 10802
    No | 5342 | 4209 | 9551

OUTCOME MEASURES:

1. Primary Outcome: Identification of a Goals of Care Conversation in the Electronic Health Record (EHR) During the Index Hospitalization
Description: Any documentation of a discussion pertaining to limitations of life sustaining treatment, palliative care, hospice, goals of care, time-limited trial, or surrogate decision makers.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | ACP Educator Led, Video Assisted Discussion | Usual Care
Number analyzed (Participants) | 6023 | 4779
Participants | 3744 | 2396

2. Secondary Outcome: Change in Documentation of Medical Orders for Resuscitation Preferences in EHR
Description: Medical records were reviewed for the presence and content of resuscitation and treatment preferences including: Full code, do not resuscitate (DNR), do not intubate (DNI), do not hospitalize (DNH), and documented preferences around feeding tubes, and dialysis. Change is measured as the number of patients with a new documented preference between baseline and 12 months.
Time Frame: Baseline, 12 months
Population: There was unanticipated high variability between receiving the intervention and the caregiver survey. Furthermore, a majority of the participants in the caregiver survey did not have any contact with the intervention at all. Accordingly, the survey activity was implemented in a fashion that did not reflect the intervention.
Measure: Number; unit: count of documentation preferences
Arm/Group | ACP Educator Led, Video Assisted Discussion | Usual Care
Number analyzed (Participants) | 6023 | 4779
count of documentation preferences
  Goals Conversation: number analyzed (Participants) | 4779 | 4779
  Goals Conversation | 3562 | 2258
  Limitation of life-sustaining treatment: number analyzed (Participants) | 4779 | 4779
  Limitation of life-sustaining treatment | 1979 | 1242
  Palliative care | 2067 | 700
  Hospice | 597 | 461
  Time-limited trials | 105 | 20
  Missing | 0 | 98

3. Secondary Outcome: Caregiver Knowledge of ACP at 12 Months
Description: 6 investigator designed questions to assess subject's knowledge of advance care planning, scores range 0-6, higher scores indicate greater knowledge
Time Frame: Baseline, 12 months
Population: There were unanticipated high variability between receiving the intervention and the caregiver survey. Furthermore, many of the participants in the caregiver survey did have any contact with the intervention at all. Accordingly, the survey activity was implemented in a fashion that did not reflect the intervention.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Groups:
- Usual Care (Control): Subjects in this arm do not meet with ACP Educator during their index hospitalization.
Arm/Group | ACP Educator Led, Video Assisted Discussion | Usual Care (Control)
Number analyzed (Participants) | 178 | 194
score on a scale | 4 [3 to 5] | 4 [3 to 5]

4. Secondary Outcome: Caregiver Confidence at 12 Months
Description: 3 investigator designed questions with responses on a 5-point likert scale from lowest to highest confidence. Range of scores 3-15, higher scores are associated with more caregiver confidence.
Time Frame: Baseline, 12 months
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | ACP Educator Led, Video Assisted Discussion | Usual Care
Number analyzed (Participants) | 178 | 194
score on a scale | 15 [10 to 15] | 15 [9 to 15]

5. Secondary Outcome: Caregiver Communication Satisfaction at 12 Months
Description: 10 investigator designed questions to assess subject's satisfaction with clinician communication. Scores range from 0-10 with higher scores indicating higher confidence. Range of scores 10-100, higher scores are associated with more satisfaction with clinician communication.
Time Frame: Baseline, 12 months
Population: as for outcome 3
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | ACP Educator Led, Video Assisted Discussion | Usual Care (Control)
Number analyzed (Participants) | 178 | 194
score on a scale | 31 [27 to 32] | 31 [26 to 32]

6. Secondary Outcome: Caregiver Decisional Satisfaction at 12 Months
Description: 12 investigator designed questions with responses on a 5-point likert scale from lowest to highest satisfaction. Range of scores 12-60, higher scores are associated with more decisional satisfaction.
Time Frame: Baseline, 12 months
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | ACP Educator Led, Video Assisted Discussion | Usual Care (Control)
Number analyzed (Participants) | 178 | 194
score on a scale | 40 [33 to 42] | 40 [36 to 43]

7. Secondary Outcome: Caregiver Decisional Certainty
Description: 2 investigator designed questions to assess level of certainty in decisions, scores range from 0-4 with highest scores indicating the highest certainty. Range of scores 0-8, higher scores are associated with more decisional certainty.
Time Frame: Baseline, 12 months
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | ACP Educator Led, Video Assisted Discussion | Usual Care (Control)
Number analyzed (Participants) | 178 | 194
score on a scale | 2 [2 to 2] | 2 [2 to 2]

ADVERSE EVENTS:
Time Frame: Adverse events were not collected because ACP is a standard part of clinical care for patients.
Description: Adverse events were not collected because ACP is a standard part of clinical care for patients.
Arm/Group | ACP Educator Led, Video Assisted Discussion | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Stepped-wedge designs have significant limitation (partial confounding by time) and should be used sparingly. Second, we looked at GOC documentation rates during index hospitalization, long-term studies looking at care delivery suggests a shard decision-making encounter. Third, we did not analyze the quality of GOC documentation during the intervention and the usual care phases.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT04857060/Prot_SAP_000.pdf